CLINICAL TRIAL: NCT02447276
Title: A Randomized, Double-Blind, Multi-Dose, Placebo-Controlled Study to Evaluate the Efficacy and Safety of REGN475 in Patients With Pain Due to Osteoarthritis of the Knee or Hip
Brief Title: Study of REGN475 in Patients With Pain Due to Osteoarthritis of the Knee or Hip
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R475-PN-1227
Record Dates: First submitted 2015-05-14; First posted 2015-05-18 (Estimated); Last update posted 2017-03-27 (Actual); Status verified 2016-10

CONDITIONS: Osteoarthritis, Knee; Osteoarthritis, Hip
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis, Hip | interventions — fasinumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Group A (Experimental): Group A will receive REGN475 dosing regimen 1
  Interventions: Drug: REGN475
- Group B (Experimental): Group B will receive REGN475 dosing regimen 2
  Interventions: Drug: REGN475
- Group C (Experimental): Group C will receive REGN475 dosing regimen 3
  Interventions: Drug: REGN475
- Group D (Experimental): Group D will receive REGN475 dosing regimen 4
  Interventions: Drug: REGN475
- Group E (Experimental): Group E will receive matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: REGN475
  Arms: Group A; Group B; Group C; Group D
Drug: Placebo
  Arms: Group E

SUMMARY:
The primary objective of this study is to evaluate the effectiveness of REGN475 compared to placebo in participants with pain due to osteoarthritis (OA) of the knee or hip and a history of inadequate joint pain relief or intolerance to current analgesic therapy.

ELIGIBILITY:
Key Inclusion Criteria:

1. Body mass index ≤39
2. Clinical diagnosis of OA of the knee or hip
3. History of inadequate pain relief or intolerance to analgesics used for OA
4. Moderate to severe pain in the index joint
5. History of regular use of analgesic medications for OA pain
6. Willing to discontinue current non-steroidal anti-inflammatory drug (NSAID) and opioid pain medications

Key Exclusion Criteria:

1. Other diseases that may involve index knee or hip, including inflammatory joint diseases, crystalline disease (gout or pseudogout), endocrinopathies, metabolic joint disease, lupus erythematosus, rheumatoid arthritis, joint infections, neuropathic disorders, avascular necrosis, Paget's disease, renal osteodystrophy or tumors
2. History of osteonecrosis, destructive arthropathy (RPOA), hip dislocation, pathologic fractures, neuropathic joint arthropathy, knee dislocation or hip dislocation
3. Trauma to the index joint in the 30 days before screening
4. Active fibromyalgia, regional pain caused by lumbar or cervical compression with radiculopathy or other moderate to severe pain that may confound assessments or self-evaluation of the pain associated with OA
5. Prior to the start of the study has received a recommendation for, or is scheduled for joint replacement surgery to be performed during the study period
6. Presence of subchondral insufficiency fracture on screening films or MRI
7. Received an intra-articular injection of hyaluronic acid in the affected index joint within 90 days prior to the screening visit
8. Systemic (ie, oral or intramuscular) corticosteroids within 30 days prior to the screening visit. Intra-articular corticosteroids in the index joint within 12 weeks of the screening visit, or to any other joint within 30 days prior to the screening visit.
9. History of autonomic neuropathy, diabetic neuropathy, or presence of clinically relevant peripheral neuropathy at the time of screening
10. Women of childbearing potential who have a positive pregnancy test result, or who do not have their pregnancy test results at baseline
11. Pregnant or breastfeeding women

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 421 (Actual)
Dates: Start 2015-05; Primary Completion 2016-03 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
The primary endpoint in the study is the change from baseline to week 16 in the Western Ontario and McMaster Osteoarthritis Index (WOMAC) pain subscale score. | Baseline to week 16

SECONDARY OUTCOMES:
Change from baseline to week 16 in the WOMAC physical function subscale score | Baseline to week 16
Change from baseline to week 16 in the Patient Global Assessment score | Baseline to week 16
Incidence of treatment-emergent adverse events (TEAEs) | Baseline to week 36 (end of study)
Incidence of anti-REGN475 antibody development | Baseline to week 36 (end of study)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (72):
- United States (72):
  - Birmingham, Alabama
  - Mobile, Alabama
  - Chandler, Arizona
  - Phoenix, Arizona
  - Tuscon, Arizona
  - Hot Spring, Arkansas
  - Little Rock, Arkansas
  - Anaheim, California
  - Beverly Hills, California
  - El Cajon, California
  - Sacramento, California
  - San Diego, California
  - Santa Ana, California
  - Thousand Oaks, California
  - Upland, California
  - Walnut Creek, California
  - Lakewood, Colorado
  - Clearwater, Florida
  - Fleming Island, Florida
  - Jacksonville, Florida
  - Miami, Florida
  - Orlando, Florida
  - Palm Harbor, Florida
  - Tamarac, Florida
  - Tampa, Florida
  - West Palm Beach, Florida
  - Weston, Florida
  - Winter Haven, Florida
  - Decatur, Georgia
  - Honolulu, Hawaii
  - Chicago, Illinois
  - Indianapolis, Indiana
  - New Orleans, Louisiana
  - Elkridge, Maryland
  - Frederick, Maryland
  - Worcester, Massachusetts
  - Saint Clair Shores, Michigan
  - Traverse City, Michigan
  - Hattiesburg, Mississippi
  - Kansas City, Missouri
  - St Louis, Missouri
  - Omaha, Nebraska
  - Brooklyn, New York
  - Hartsdale, New York
  - New York, New York
  - Plainview, New York
  - Rochester, New York
  - Charlotte, North Carolina
  - High Point, North Carolina
  - Raleigh, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Oklahoma City, Oklahoma
  - Tulsa, Oklahoma
  - Bensalem, Pennsylvania
  - Duncansville, Pennsylvania
  - Jenkintown, Pennsylvania
  - Warwick, Rhode Island
  - Mt. Pleasant, South Carolina
  - Jackson, Tennessee
  - Jefferson City, Tennessee
  - Memphis, Tennessee
  - Cypress, Texas
  - Dallas, Texas
  - Lubbock, Texas
  - Mesquite, Texas
  - Plano, Texas
  - Waco, Texas
  - Salt Lake City, Utah
  - Sandy City, Utah
  - West Jordan, Utah
  - Norfolk, Virginia

REFERENCES:
- [Derived] Eng S, Fetell M, Gao H, Mei J, Trejos J, Cortes-Burgos L, Ho T, Manvelian G, Patel Y, Trinh N, Turner KC, Hassan HE, DiMartino S, Krueger P, Geba GP, Braunstein N, Macdonald LE, Soltys R, Croll SD, Dakin P. The Effects of Fasinumab on Peripheral Nerve Function and Ganglion Anatomy: Results From a Randomized, Double-Blind, Placebo-Controlled Study in Patients With Pain Due to Osteoarthritis of the Knee or Hip, and a Series of Nonclinical Studies. Curr Ther Res Clin Exp. 2025 Oct 24;103:100813. doi: 10.1016/j.curtheres.2025.100813. eCollection 2025. PMID 41323020
- [Derived] Dakin P, DiMartino SJ, Gao H, Maloney J, Kivitz AJ, Schnitzer TJ, Stahl N, Yancopoulos GD, Geba GP. The Efficacy, Tolerability, and Joint Safety of Fasinumab in Osteoarthritis Pain: A Phase IIb/III Double-Blind, Placebo-Controlled, Randomized Clinical Trial. Arthritis Rheumatol. 2019 Nov;71(11):1824-1834. doi: 10.1002/art.41012. Epub 2019 Sep 20. PMID 31207169